CLINICAL TRIAL: NCT03452267
Title: Effect of Metformin and Pioglitazone on Insulin Signaling in Skeletal Muscle
Brief Title: Insulin Signaling in Skeletal Muscle
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Kyle Jon Burghardt, Pharm.D., Assistant Professor of Pharmacy Practice, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MetPioMuscle
Record Dates: First submitted 2018-02-12; First posted 2018-03-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — oral, 850 mg twice daily
  Arms: Metformin
Drug: Pioglitazone — oral, 45 mg daily
  Arms: Pioglitazone
Drug: Placebo — oral, once daily
  Arms: Placebo

SUMMARY:
The insulin sensitizing effects of metformin and pioglitazone in the skeletal muscle remain unknown. Our group aims to analyze molecular changes within the skeletal muscle of pre-diabetic patients through the use of a clinical trial in humans.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes as defined by an oral glucose tolerance test 2-hour level between 140 and 200 mg/dL

General Inclusion Criteria:

* Able to communicate meaningfully with the investigator and legally competent to provide informed written consent.
* Female subjects must be non-lactating, have a negative pregnancy test, and be on acceptable birth control.

Exclusion Criteria:

* Oral glucose tolerance test <140 or >200mg/dL
* Treated with any of the following medications:

  * Systemic glucocorticoids (more than 2 weeks), antineoplastic agents, transplant medications, fibrates, anti-retroviral medications, or thiazolidinediones within 6 months prior to screening
  * Start or change of hormonal replacement therapy within 3 months prior to screening
  * Short-acting insulin (more than15 units per day) in DMT2 subjects, indicating severe insulin deficiency within 6 months prior to screening
* History or presence of any of the following conditions:

  * Clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG)
  * Peripheral vascular disease (history of claudication)
  * Clinically significant pulmonary disease.
  * Current uncontrolled hypertension (systolic BP>160 mmHg, diastolic BP>100 mmHg)
  * History or presence of malignancy other than basal cell or squamous cell skin cancer
  * Autonomic neuropathy
  * Clinically significant hematologic disease
* Any of the following abnormal laboratory values:

  * Hematocrit < 35 vol%
  * Serum creatinine > 1.6 mg/dl
  * AST, ALT or Alkaline phosphatase > 2.5 times the upper limit of normal
  * PT, PTT outside the normal reference range
  * TSH outside the normal reference range
  * Triglycerides > 400 mg/dl
  * Platelet count < 50,000
* Current or history of drug abuse or alcohol abuse
* Blood donation within 2 months prior to screening
* Engage in exercise with moderate to hard intensity for greater than 1 hour per day for 5 or more days per week.
* Diagnosed with Type 1 diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proteomic | 3 months
  Changes in global protein abundance levels
Proteomic 2 | 3 months
  Changes in global protein phosphorylation levels

SECONDARY OUTCOMES:
Epigenomic | 3 months
  Change in global DNA percent methylation

IPD SHARING:
Plan to Share IPD: No